CLINICAL TRIAL: NCT00357643
Title: Effect of Calcium and Vitamin D on Bone Loss From the Hip
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tufts University (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U01AG010353 (NIH)
Record Dates: First submitted 2006-07-26; First posted 2006-07-27 (Estimated); Last update posted 2006-07-27 (Estimated); Status verified 2005-06

CONDITIONS: Osteoporosis
Keywords: calcium; vitamin D; bone loss
MeSH Terms: conditions — Osteoporosis; Bone Diseases, Metabolic | interventions — Calcium; Vitamin D

INTERVENTIONS:
Drug: Calcium 500 mg/day and vitamin D 700 IU/day

SUMMARY:
The primary aim of this study is to determine the effects of supplementation with both calcium and vitamin D on changes in bone density of the hip in men and women age 65 and older.

DETAILED DESCRIPTION:
In this study 445 men and women age 65 and older were enrolled for three years each. Subjects were randomized to treatment with 500 mg of calcium s calcium citrate malate plus 700 IU of vitamin D daily or placebo. Subjects came to the research center every six months for biochemical and bone mineral density measurements. Changes in these measures over the three years were determined in each group and compared.

ELIGIBILITY:
Inclusion Criteria:

>65 years calcium intake < 1500 mg/day Willing to discontinue calcium and vitamin D pills for 2 months prior to enrollment

Exclusion Criteria:

Mentally incompetent, femoral neck BMD greater than 2 SD above/below age/sex-matched reference mean, 24-hr urine calcium/creatinine > 300 mg/d women or >350 mg/d men terminal illness, renal disease requiring treatment, kidney stone in the past 10 years, current hyperparathyroidism, treated with glucocorticoids, estrogen or androgen, fluoride, calcitonin, bisphosphonate, or any other treatment for osteoporosis.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 450
Dates: Start 1992-10; Study Completion 1996-02

PRIMARY OUTCOMES:
Bone Density of the hip

SECONDARY OUTCOMES:
Annual and Seasonal patterns of change in bone mineral density of the hip
Associations between biochemical, physical and life-style factors
Examine influence of clinical status, lifestyle, medication use and season on the occurrence of falls

CONTACTS AND LOCATIONS:
Overall Officials: Bess Dawson-Hughes, MD, Principal Investigator — Tufts University
Locations (1):
- Human Nutrition Research Center on Aging at Tufts U, Boston, Massachusetts, United States

REFERENCES:
- [Result] Dawson-Hughes B, Harris SS, Krall EA, Dallal GE. Effect of calcium and vitamin D supplementation on bone density in men and women 65 years of age or older. N Engl J Med. 1997 Sep 4;337(10):670-6. doi: 10.1056/NEJM199709043371003. PMID 9278463
- [Derived] Dawson-Hughes B, Harris SS, Ceglia L, Palermo NJ. Serum sclerostin levels vary with season. J Clin Endocrinol Metab. 2014 Jan;99(1):E149-52. doi: 10.1210/jc.2013-3148. Epub 2013 Dec 20. PMID 24248178
- [Derived] Pittas AG, Harris SS, Stark PC, Dawson-Hughes B. The effects of calcium and vitamin D supplementation on blood glucose and markers of inflammation in nondiabetic adults. Diabetes Care. 2007 Apr;30(4):980-6. doi: 10.2337/dc06-1994. Epub 2007 Feb 2. PMID 17277040